CLINICAL TRIAL: NCT07066228
Title: Clinical Transformation of Bone Reconstruction With Autologous Bone Marrow Mesenchymal Stem Cells in Vitro to Repair Long Tubular Bone Defects of Limbs
Brief Title: Bone Reconstruction With Autologous Bone Marrow Mesenchymal Stem Cells in Vitro to Repair Long Tubular Bone Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEBLTBD-2022-02
Record Dates: First submitted 2025-04-11; First posted 2025-07-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Defective Composite Restorations; Bone Cysts; Bone Defect; Bone Nonunion
Keywords: autologous bone marrow mesenchymal stem cells; DBM; long tubular bone defects of limbs
MeSH Terms: conditions — Bone Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tissue engineered bone on bone defect (Other)
  Interventions: Device: tissue-engineered bone

INTERVENTIONS:
Device: tissue-engineered bone — Commercial decalcified bone scaffolds were combined with autologous bone marrow mesenchymal stem cells to form tissue engineered bone in vitro

SUMMARY:
Commercial decalcified bone scaffolds were combined with autologous bone marrow mesenchymal stem cells to form tissue engineered bone in vitro to explore the effect of this tissue engineered bone in the clinical repair of long tubular bone defects in limbs.

DETAILED DESCRIPTION:
Bone defects caused by trauma, tumors, and other factors, particularly weight-bearing long tubular bone defects in the limbs, pose significant harm to patients and severely impact their quality of life, remaining a major clinical challenge. Current repair methods such as autologous bone grafting, vascularized autologous bone grafting, allogeneic bone grafting, induced membrane technique, and bone transport technique face limitations including lengthy treatment cycles, high costs, restricted donor sites and bone harvest quantities, and unpredictable outcomes.

To address these challenges, the National Engineering Research Center for Tissue Engineering has developed an innovative approach through continuous research and innovation. This method utilizes autologous bone marrow mesenchymal stem cells (BMSCs) with minimal invasiveness, strong proliferation capacity, and potent osteogenic potential as seed cells for bone construction. These cells are combined with clinically approved allogeneic decalcified bone materials to create tissue-engineered bone through in vitro induction. This approach offers multiple advantages: absence of immune rejection, unrestricted material sources, sufficient cultured bone volume, and high survival rates, providing a new direction for treating long tubular bone defects in limbs.

This study aims to evaluate the clinical efficacy of tissue-engineered bone constructed with autologous BMSCs for repairing long bone defects in extremities, thereby providing evidence-based support for bone defect treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-55 years old, gender unrestricted;
2. Defective nonunion with bone loss exceeding 30% of the bone cross-section and a length of 2-3 cm;
3. Solitary bone cysts involving more than 50% of the bone cross-section.

Exclusion Criteria:

1. Combined with local tumors, tuberculosis, infections or other bone-healing affecting lesions;
2. Systemic diseases affecting bone healing such as osteofibrous dysplasia, osteogenesis imperfecta, bone dystrophic diseases, and metabolic bone disorders;
3. Moderate-to-severe osteoporosis (BMD: T-score < -2.5);
4. Severe systemic conditions including systemic malnutrition, systemic infectious diseases, severe cardiopulmonary diseases, coagulation disorders, and major organ failure;
5. Complicated with severe brain trauma;
6. Heavy smoking, drug abuse, alcoholism, or other harmful addictions;
7. Psychiatric disorders or patients with menopausal symptoms;
8. Concurrent participation in other studies or recent completion (within 4 weeks) of other clinical trials;
9. Pregnancy, lactation, or planned pregnancy within one year after initial enrollment;
10. Psychological conditions impairing treatment compliance;
11. Congenital malformations of vital organs or other systems;
12. Nonunion caused by malignant tumor resection;
13. Refusal to accept tissue-engineered bone repair protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The scores of bone healing | About 360 days after surgical treatment of bone defect
  The scores of bone healing are divided into three kinds: nonhealing: 0；delayed healing: 1; normal healing.
The adverse event incidence using tissue-engineered bone | About 360 days after surgical treatment of bone defect
  The adverse event incidence of tissue-engineered bone
Bone union (bone healing) evaluation through modified lane and sandhu radiological scoring system | At the end of visits 1, 2, 3 (respectively performed at screening and 7, 90, 360 days after the surgery)
  Evaluation of the bone regeneration in the area of intervention in comparison to baseline (V1), by means of X-ray and/or CT scan examination, on visits V1, V2 and V3. X-ray scoring systems have been implemented according to the criteria proposed by modified Lane and Sandhu Radiological Scoring System. This scoring system evaluates bone formation and union. To evaluate the bone formation, there is a scale with 5 points, from 0 to 4 (0=No evidence of bone formation-4=Bone formation occupying 100% of defect). To evaluate bone union, there is a scale with 3 points, from 0 to 2 (0=Non-union-2=Radiogrical union)

SECONDARY OUTCOMES:
The scores of time of weight loading after operation | About 360 days after surgical treatment of bone defect
  The scores of time of weight loading after operation are divided into three kinds: longer than six months: 0; longer than three months: 1; less than three months: 2
The scores of pain | About 360 days after surgical treatment of bone defect
  The scores of pain after operation are divided into four kinds: severe: 0; moderate: 1; slight: 2; none: 3.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Ren, Principal Investigator — The First Affiliated Hospital of Xinxiang Medical College
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China